CLINICAL TRIAL: NCT03140553
Title: TCH (Docetaxel/Carboplatin/Trastuzumab) Versus EC -TH(Epirubicin/Cyclophosphamide Followed by Docetaxe/Trastuzumab) as Neoadjuvant Treatment for HER2-Positive Breast Cancer
Brief Title: TCH Versus EC-TH as Neoadjuvant Treatment for HER2-Positive Breast Cancer
Acronym: neoCARH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, KunWang, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170308
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: HER2-Positive Breast Cancer
Keywords: Neoadjuvant Treatment; HER2-Positive Breast Cancer
MeSH Terms: interventions — Docetaxel; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCH (Experimental): docetaxel/carboplatin/trastuzumab
  Interventions: Drug: TCH (docetaxel/carboplatin/trastuzumab) versus EC-TH(epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab)
- EC-TH (Active Comparator): epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab
  Interventions: Drug: TCH (docetaxel/carboplatin/trastuzumab) versus EC-TH(epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab)

INTERVENTIONS:
Drug: TCH (docetaxel/carboplatin/trastuzumab) versus EC-TH(epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab) — TCH (docetaxel/carboplatin/trastuzumab) versus EC followed by TH(epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab) as Neoadjuvant Treatment for HER2-Positive Breast Cancer

SUMMARY:
Both TCH (docetaxel/carboplatin/trastuzumab) and EC followed by TH(epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab) regimens as Neoadjuvant Treatment for HER2-Positive Breast Cancer have been recommended by NCCN guideline. It is unknown which regimen is better. This study is to evaluate the efficacy and safety of TCH (docetaxel/carboplatin/trastuzumab) and EC followed by TH(epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab) regimens as Neoadjuvant Treatment in HER2-Positive breast cancer. The endpoint of pathologic complete response is used as a surrogate marker for survival. Safety and tolerability assessed by number of grade 4 toxicities and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HER2 positive invasive breast carcinoma
* Clinical stage Ⅱ-ⅢC
* Eastern Cooperative Oncology Group(ECOG) performance status 0 to 1 within 14 days of study entry
* Normal (greater than 50%) left ventricular ejection fraction (LVEF) by echocardiography
* Signed informed consent
* Adequate organ function within 2 weeks of study entry:

Absolute neutrophil count >1500/mm3, Hgb >9.0 g/dl and platelet count >100,000/mm3 Total bilirubin < upper limit of normal Creatinine < 1.5 mg/dL or calculated cranial cruciate ligament (CrCL) >50mL/min using the Cockcroft Gault equation serum glutamate oxaloacetate transaminase(SGOT)(AST) or serum glutamic oxaloacetic transaminase(SGPT)(ALT) and Alkaline Phosphatase must be within the range allowing for eligibility

* Patients must be over 18 years old.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Metastatic disease
* Prior chemotherapy, hormonal therapy, biologic therapy, investigational agent, targeted therapy or radiation therapy for current breast cancer. Patients with history of breast cancer greater than 5 years from initial diagnosis are eligible for the study. Patients may not have received anthracycline-based chemotherapy in the past. Patients with history of ductal carcinoma in situ(DCIS) are eligible if there were treated with surgery alone.
* History of previous or current malignancy at other sites with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies, who remain disease free for greater than five years are eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
pCR | one year
  pathologic complete response

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yang C, Li P, Chen Y, Zheng J, Zhang X, Gao HF, Zhang L, Wang K. Pooled analysis of NeoCARH and NeoCART trials: patient-reported outcomes in patients with early-stage breast cancer receiving platinum-based or anthracycline-based neoadjuvant chemotherapy. Support Care Cancer. 2024 Jun 3;32(6):401. doi: 10.1007/s00520-024-08610-3. PMID 38829506
- [Derived] Gao HF, Wu Z, Lin Y, Song XY, Cao Y, Chen QJ, Zhang G, Fu P, Liu Z, Zhang LL, Yang CQ, Yang M, Zhu T, Ji F, Li JQ, Cheng MY, Wang K. Anthracycline-containing versus carboplatin-containing neoadjuvant chemotherapy in combination with trastuzumab for HER2-positive breast cancer: the neoCARH phase II randomized clinical trial. Ther Adv Med Oncol. 2021 Apr 20;13:17588359211009003. doi: 10.1177/17588359211009003. eCollection 2021. PMID 33959195
- [Derived] Li WP, Zhu T, Hu MX, Yang M, Ji F, Gao HF, Yang CQ, Zhang LL, Cheng MY, Xu FP, Wang K. Comparison of the efficacy and safety of the EC-T (epirubicin/cyclophosphamide followed by docetaxel) and TCb (docetaxel/carboplatin) neoadjuvant regimens in early TOP2A-normal stage II-III breast cancer. Neoplasma. 2020 Nov;67(6):1409-1415. doi: 10.4149/neo_2020_200130N96. Epub 2020 Jul 13. PMID 32657611